CLINICAL TRIAL: NCT06520423
Title: Effectiveness of Urethral Stent Irrigation in Preventing Surgical Site Infections in Adolescents With Hypospadias: A Multicenter Randomized Controlled Trial
Brief Title: Effectiveness of Urethral Stent Irrigation in Preventing Surgical Site Infections in Adolescents With Hypospadias
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xing Liu (Other)
Responsible Party: Sponsor-Investigator, Xing Liu, Professor, Doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024258
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two intervention arms. A computer-generated randomization sequence-created by staff not involved in trial execution or analysis-will ensure allocation concealment. Assignments will be sealed in sequentially numbered, opaque envelopes held by a clinician independent of the study team.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary catheter drainage (Active Comparator): These patients will undergo urinary catheter drainage for seven days following urethroplasty
  Interventions: Procedure: Urinary catheter drainage
- Urethral stent tube irrigation (combined with urinary catheter drainage) (Experimental): These patients will undergo urinary catheter drainage (combined with urinary catheter drainage) for seven days following urethroplasty
  Interventions: Procedure: Urethral stent tube irrigation; Procedure: Urinary catheter drainage

INTERVENTIONS:
Procedure: Urethral stent tube irrigation — During urethroplasty, a Fr3 ureteral catheter will be placed in the reconstructed urethra, with the proximal end extending approximately 2 cm beyond the urethral wound. The distal end will connect to an F6 single-lumen ureter and a urinary bag. On the second postoperative day, the urethra will be irrigated with 5 ml of saline twice daily. This irrigation routine will continue until the catheter is removed.
  Arms: Urethral stent tube irrigation (combined with urinary catheter drainage)
Procedure: Urinary catheter drainage — During urethroplasty, intraurethral retention of urethral catheters is used to drain urine from the bladder.

SUMMARY:
This multicenter randomized controlled trial aims to determine whether urethral stent tube irrigation, combined with urinary catheter drainage, prevents postoperative wound infections compared to urinary catheter drainage alone in adolescents with hypospadias.

DETAILED DESCRIPTION:
Hypospadias is one of the most common genital developmental malformations in pediatric patients, with a prevalence of approximately 0.5%. The primary manifestations of hypospadias include an ectopic urethral opening, penile recurvature, and abnormal distribution of the prepuce. Currently, urethroplasty is the only treatment for hypospadias, with surgery recommended within the first three years of life. However, due to economic, cultural, and social factors, many children miss the optimal age for surgery and require initial or re-repair surgery during puberty. Additionally, some children who underwent hypospadias repair before puberty develop penile recurvature and other complications during adolescence, necessitating reoperation. Physiological changes during puberty, such as penile growth, pubic hair development, increased skin appendages, secretions, and frequency of erections, increase the risk of wound infection and poor healing post-surgery. To address these issues, we placed a stent in the reconstructed urethra of adolescents with hypospadias and performed urethral irrigation postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with hypospadias and in Tanner stages II-V at the Department of Urology, Affiliated Children's Hospital of Chongqing Medical University.
2. Patients and their guardians have been informed about the nature of the study, understand the protocol, can ensure compliance, and have signed an informed consent form.

Exclusion Criteria:

1. Patients undergoing meatal advancement and glanuloplasty (MAGPI) only.
2. Patients undergoing penile recurvature correction only.
3. Patients undergoing only urethral fistula formation/urethrostomy.
4. Patients with a prostatic utricle.
5. Patients with contraindications to the procedure, such as severe cardiac disease, systemic or localized infection, thrombocytopenia, coagulation disorders, congenital immunodeficiencies, or uncontrolled diabetes mellitus.
6. Patients already enrolled in or during the follow-up of other clinical studies. Patients who do not wish to participate in this study or demonstrate poor compliance with follow-up requirements.

Ages: 9 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Overall complication rate | 12 months
  Probability of overall complications following urethroplasty in adolescent boys with hypospadias.
Specific complication rates | 12 months
  Probability of specific complications following urethroplasty in adolescent boys with hypospadias.

SECONDARY OUTCOMES:
Urinary function | 12 months
  Urinary function was evaluated using non-validated questions addressing urinary stream, urinary power, the presence of post-void dribbling, and straining during voiding. Urinary function outcomes were assessed using patient-reported categorical and ordinal measures (urinary stream pattern, urinary power, post-void dribbling, and straining), rather than a composite scoring scale; therefore, no minimum or maximum scale values apply. For ordinal outcomes, higher categories indicate worse urinary symptoms.
Cosmetic outcomes | 12 months
  Cosmetic outcomes were assessed using the Pediatric Penile Perception Score (PPPS), a 4-point ordinal scale ranging from 1 (very dissatisfied) to 4 (very satisfied), with higher scores indicating better cosmetic outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Liu, Doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Apart from the participant's personal information.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: Apart from the participant's personal information.

REFERENCES:
- [Background] Lund L, Engebjerg MC, Pedersen L, Ehrenstein V, Norgaard M, Sorensen HT. Prevalence of hypospadias in Danish boys: a longitudinal study, 1977-2005. Eur Urol. 2009 May;55(5):1022-6. doi: 10.1016/j.eururo.2009.01.005. Epub 2009 Jan 13. PMID 19155122
- [Background] Weber DM, Schonbucher VB, Gobet R, Gerber A, Landolt MA. Is there an ideal age for hypospadias repair? A pilot study. J Pediatr Urol. 2009 Oct;5(5):345-50. doi: 10.1016/j.jpurol.2008.12.008. Epub 2009 Jan 30. PMID 19186110
- [Background] Marshall WA, Tanner JM. Variations in the pattern of pubertal changes in boys. Arch Dis Child. 1970 Feb;45(239):13-23. doi: 10.1136/adc.45.239.13. PMID 5440182
- [Background] Zheng DC, Wang H, Lu MJ, Chen Q, Chen YB, Ren XM, Yao HJ, Xu MX, Zhang K, Cai ZK, Wang Z. A comparative study of the use of a transverse preputial island flap (the Duckett technique) to treat primary and secondary hypospadias in older Chinese patients with severe chordee. World J Urol. 2013 Aug;31(4):965-9. doi: 10.1007/s00345-012-0990-2. Epub 2012 Nov 23. PMID 23179731
- [Background] Hensle TW, Tennenbaum SY, Reiley EA, Pollard J. Hypospadias repair in adults: adventures and misadventures. J Urol. 2001 Jan;165(1):77-9. doi: 10.1097/00005392-200101000-00019. PMID 11125368
- [Background] Cakmak M, Caglayan F, Kilic D, Kaygusuz S, Cakmak A, Ulusoy S, Ozlu N, Ozluk O. Efficacy of povidone-iodine in preputial antisepsis. Int J Clin Pract. 2003 Nov;57(9):752-4. PMID 14686562
- [Background] Li LC, Zhang X, Zhou SW, Zhou XC, Yang WM, Zhang YS. Experience with repair of hypospadias using bladder mucosa in adolescents and adults. J Urol. 1995 Apr;153(4):1117-9. PMID 7869477